CLINICAL TRIAL: NCT04565249
Title: A Randomized, Double-blind, Dose-ranging, Placebo Controlled, Phase 2a Evaluation of the Safety, Tolerability, and Pharmacokinetics of PLN-74809 in Participants With Acute Respiratory Distress Syndrome (ARDS) Associated With at Least Severe COVID-19 (INTEGRIS-ARDS)
Brief Title: Evaluation of the Safety, Tolerability, and Pharmacokinetics of PLN-74809 in Participants With Acute Respiratory Distress Syndrome (ARDS) Associated With at Least Severe COVID-19
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study halted and will not resume; participants are no longer being examined or receiving intervention
Sponsor: Pliant Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PLN-74809-ARDS-204
Record Dates: First submitted 2020-09-15; First posted 2020-09-25 (Actual); Results first posted 2022-11-17 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2020-09

CONDITIONS: Acute Respiratory Distress Syndrome; SARS-CoV-2
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- PLN-74809 Dose Level1 (Experimental): Dose Level 1 of PLN-74809
  Interventions: Drug: PLN-74809; Drug: Placebo
- PLN-74809 Dose Level 2 (Experimental): Dose Level 2 of PLN-74809
  Interventions: Drug: PLN-74809; Drug: Placebo
- PLN74809 Dose Level 3 (Experimental): Dose Level 3 of PLN-74809
  Interventions: Drug: PLN-74809; Drug: Placebo

INTERVENTIONS:
Drug: PLN-74809 — PLN-74809
Drug: Placebo — Placebo

SUMMARY:
Evaluation of the safety, tolerability, and pharmacokinetics of PLN-74809 in participants with acute respiratory distress syndrome (ARDS) associated with at least severe COVID-19

DETAILED DESCRIPTION:
Approximately 36 participants will be enrolled sequentially into 3 cohorts. Within each cohort of 12 participants, 9 will be randomized to PLN-74809 and 3 will be randomized to placebo (3:1 ratio).

* In Part 1, approximately 12 participants will be randomized to Dose level 1 of PLN-74809 or placebo QD
* In Part 2, approximately 12 participants will be randomized to Dose level 2 of PLN-74809 or placebo QD
* In Part 3, approximately 12 participants will be randomized to Dose level 3 of PLN-74809 or placebo QD

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ARDS (Berlin Criteria)
* Hospitalized with at least severe COVID-19 (FDA 2020)
* Receiving support for acute lung injury/respiratory distress via supplemental oxygen
* Serum aspartate aminotransferase (AST) concentration ≤ 120 U/L and serum alanine aminotransferase (ALT) concentration ≤ 150 U/L
* Serum total bilirubin ≤ 1.8 mg/dL, in the absence of Gilbert's syndrome or hemolysis

Exclusion Criteria:

* Greater than 72 hours since time of onset of ARDS.
* Greater than 7 days since start of mechanical ventilation.
* Currently receiving or anticipated to receive extracorporeal life support (ECLS), extracorporeal membrane oxygenation (ECMO) or high-frequency oscillatory ventilation
* Unwillingness to follow lung protective ventilation strategy (i.e., tidal volume of 6 mL/kg of predicted body weight and prone positioning) and fluid management protocol (Fluids and Catheters Treatment Trial [FACTT] Conservative or Lite) per local institutional standards (HFOV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pliant Therapeutics, Study Director — Pliant Therapeutics, Inc.
Locations (6):
- United States (6):
  - Valleywise Health Medical Center, Phoenix, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - National Jewish Health, Denver, Colorado
  - Advent Health, Orlando, Florida
  - Augusta University Medical Center, Augusta, Georgia
  - Atlantic Health System, Summit, New Jersey

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was discontinued prior to completion of enrollment of Dose 1 due to the lack of participant availability following the introduction of COVID-19 vaccines as well as the increased and successful measures to contain the virus leading to a dramatic decrease in the number of severe and critical COVID-19 patients with ARDS.
Groups:
- PLN-74809: Dose 1 (40 mg): N=5
- PLN-74809: Dose 2 (80 mg); PLN-74809: Dose 3 (160 mg): not enrolled (study discontinued)
- Placebo: N=1
Period: Overall Study
Arm/Group | PLN-74809: Dose 1 (40 mg) | PLN-74809: Dose 2 (80 mg) | PLN-74809: Dose 3 (160 mg) | Placebo
Started | 5 | 0 | 0 | 1
Completed | 5 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Study was discontinued before completion of enrollment of Dose 1.
Groups:
- Total: Total of all reporting groups
Arm/Group | PLN-74809: Dose 1 (40 mg) | PLN-74809: Dose 2 (80 mg) | PLN-74809: Dose 3 (160 mg) | Placebo | Total
Number analyzed (Participants) | 5 | 0 | 0 | 1 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (6.54) |  |  | 58.0 (0) | 57.5 (5.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 |  |  | 0 | 3
  Male | 2 |  |  | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  | 0 | 0
  Asian | 0 |  |  | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 |  |  | 0 | 0
  Black or African American | 1 |  |  | 0 | 1
  White | 4 |  |  | 1 | 5
  More than one race | 0 |  |  | 0 | 0
  Unknown or Not Reported | 0 |  |  | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events and Laboratory Abnormalities, Assessed by CTCAE V5.0
Description: Number of Participants With Treatment-related Adverse Events and Laboratory Abnormalities which was Assessed by CTCAE V5.
Time Frame: Adverse events were collected from the time the participant signed the Informed Consent Form until the Day 28 study visit
Population: 5 Participant received PLN-74809 and 1 participant received Placebo
Measure: Number; unit: participants
Groups:
- PLN-74809: Dose Level 1 (40 mg): N=5
- PLN-74809: Dose Level 2 (80 mg); PLN-74809: Dose Level 3 (160 mg): Not enrolled (study discontinued)
Arm/Group | PLN-74809: Dose Level 1 (40 mg) | PLN-74809: Dose Level 2 (80 mg) | PLN-74809: Dose Level 3 (160 mg) | Placebo
Number analyzed (Participants) | 5 | 0 | 0 | 1
participants | 0 |  |  | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the Informed Consent Form was completed until Day 28 study visit.
Description: No participants were enrolled in Doses 2 and 3.
Arm/Group | PLN-74809: Dose Level 1 (40 mg) | PLN-74809: Dose Level 2 (80 mg) | PLN-74809: Dose Level 3 (160 mg) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/0 | 0/0 | 1/1
Serious Adverse Events (participants affected / at risk) | 3/5 | 0/0 | 0/0 | 1/1
Other Adverse Events (participants affected / at risk) | 5/5 | 0/0 | 0/0 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLN-74809: Dose Level 1 (40 mg) (N=5) | PLN-74809: Dose Level 2 (80 mg) (N=0) | PLN-74809: Dose Level 3 (160 mg) (N=0) | Placebo (N=1)
Respiratory rate increased (Investigations) | 0 | 0 | 0 | 1
Intestinal Dilatation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal Compartment Syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ventricular Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac Arrest (Cardiac disorders) | 0 | 0 | 0 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLN-74809: Dose Level 1 (40 mg) (N=5) | PLN-74809: Dose Level 2 (80 mg) (N=0) | PLN-74809: Dose Level 3 (160 mg) (N=0) | Placebo (N=1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 | 0 | 0
Cardiac Aneurysm (Cardiac disorders) | 1 (1) | 0 | 0 | 0
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 (1) | 0 | 0 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 0 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 2 (2) | 0 | 0 | 0
Electrocardiogram QT Prolonged (Investigations) | 1 (1) | 0 | 0 | 0
Klebsiella Test Positive (Investigations) | 1 (1) | 0 | 0 | 0
Staphylococcus Test Positive (Investigations) | 1 (1) | 0 | 0 | 0
Stenotrophomonas Test Positive (Investigations) | 1 (1) | 0 | 0 | 0
Fluid Overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 | 0 | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 0 | 0
Subcutaneous Emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 0 | 0 | 0
Embolism (Vascular disorders) | 1 (1) | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 (1) | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was discontinued prior to completion of enrollment of Dose 1 due to the lack of participant availability following the introduction of COVID-19 vaccines as well as the increased and successful measures to contain the virus leading to a dramatic decrease in the number of severe and critical COVID-19 patients with ARDS. As a result, the study did not reach the target number of participants needed to achieve target power and statistically reliable results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Per protocol, the data generated in this clinical study are the exclusive property of the Sponsor and are confidential. Any publication of the results of this study must be authorized by the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2020-10-23): https://cdn.clinicaltrials.gov/large-docs/49/NCT04565249/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-13): https://cdn.clinicaltrials.gov/large-docs/49/NCT04565249/SAP_001.pdf